CLINICAL TRIAL: NCT01433809
Title: Biomarkers in Thyroid Cancer
Brief Title: Biomarkers to Distinguish Benign From Malignant Thyroid Neoplasm
Status: Completed | Type: Observational
Sponsor: Norman Eberhardt (Other)
Responsible Party: Sponsor-Investigator, Norman Eberhardt, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 11-002846
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Cancer of the Thyroid; Neoplasms, Thyroid; Thyroid Adenoma; Thyroid Cancer; Thyroid Carcinoma
Keywords: thyroid cancer; thyroid neoplasm; thyroid adenoma
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, RNA/DNA from fine needle aspirate biopsies of thyroid nodules, fresh frozen surgical tissue, formalin fixed paraffin embedded tissue.
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol will evaluate microRNA biomarkers in blood and fine-needle aspirate biopsies (FNAB) of thyroid nodules. MicroRNA profiles will be determined and evaluated for their utility in pre-operative diagnosis, in particular to distinguish benign from malignant throid neoplasms. Post-surgical fresh-frozen thyroid cancer tissue will be assessed for somatic mutations, mRNA, and microRNA expression patterns. FFPE tissue will be used to obtain H&E and unstained slides to specific biomarker results using immunohistochemistry.

DETAILED DESCRIPTION:
This protocol requires the collection of blood (5 ml), fine-needle aspirate biopsies (FNAB), and post-surgical thyroid cancer tissue. The post surgical tissue includes fresh-frozen tissue that is considered waste and in excess of that required for pathologic diagnosis, and archived formalin-fixed, paraffin-embedded tissue (FFPE). The blood will be used as a substrate for assessing known markers, including microRNA expression patterns that may be useful to predict disease and thyroid cancer morphotype. The FNABs will be used to screen the potential of markers for pre-operative diagnosis. The post-surgical fresh-frozen thyroid cancer tissue will be used to isolate DNA and RNA in order to assess somatic mutations (RAS and PAX8/PPAR-gamma rearrangement) and messenger RNA, and microRNA expression patterns. The FFPE tissue will be used to obtain H&E and unstained slides to validate results using immunohistochemistry. The goal of these studies is to define molecular markers that will accurately distinguish benign from malignant disease and the multiple thyroid cancer phenotypes. Current methods of distinguishing benign from malignant disease requires a detailed post-surgical analysis and no known markers have yet been identified to reliably differentiate the multiple thyroid cancer morphotypes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with palpable thyroid nodule suspicious for thyroid neoplasm
* Patient selected to undergo fine needle biopsy for cytologic diagnosis
* Male (18 years of age or older)
* Female (18 years of age or older)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals undergoing fine needle biopsy for diagnosis of thyroid cancer, who provide written consent to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Distinguish follicular adenoma from follicular carcinoma | 3 years
  Biomarkers will be identified to distinguish benign follicular adenoma from follicular carcinoma of the thyroid.

CONTACTS AND LOCATIONS:
Overall Officials: Norman Eberhardt, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States